CLINICAL TRIAL: NCT06987799
Title: Addressing Depression for African American Adults With Hypertension: Applying Community-Engaged Implementation Science
Brief Title: Community-based Approach to Lowering Stress Through Mindfulness
Acronym: CALM-Chicago
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Total Resource Community Development Organization (TRCDO) (Unknown)
Responsible Party: Principal Investigator, Allison Carroll, Assistant Professor, Northwestern University Feinberg School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00215977; K23HL168234 (NIH)
Record Dates: First submitted 2025-05-05; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Depression; Hypertension
Keywords: culturally adapted; african american; depression; high blood pressure; hypertension
MeSH Terms: conditions — Depression; Hypertension | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Culturally adapted mindfulness-based stress reduction intervention (Experimental): This arm will participate in the CALM-Chicago intervention, a culturally adapted mindfulness-based stress reduction intervention that has been further adapted for implementation in faith-based communities on the South Side of Chicago. The intervention includes 8 weekly group sessions in which participants receive education about mindfulness, stress reduction, and blood pressure management; practice mindfulness activities and meditation; and develop a personal mindfulness practice.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR; CALM-Chicago Study)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR; CALM-Chicago Study) — This clinical trial will evaluate the effectiveness of the culturally adapted intervention, CALM-Chicago, in a community setting. CALM-Chicago has been previously used in a clinical setting.
  Other Names: CALM-Chicago; M-Body

SUMMARY:
The goal of this clinical trial is to test a culturally adapted mindfulness-based stress reduction intervention in a community setting for African American adults with high blood pressure (hypertension) and depression. The main questions it aims to answer are:

* Does participation in a culturally adapted mindfulness-based intervention improve depressive symptoms?
* Does participation in a culturally adapted mindfulness-based intervention improve blood pressure control?
* Is the intervention acceptable, appropriate, and feasible as delivered in a community setting?

Participants will:

* Participate in an 8-week group-based mindfulness intervention (CALM-Chicago). During intervention sessions, participants will learn about mindfulness and stress management and complete mindfulness-based activities, such as guided deep breathing and meditation.
* Complete surveys online
* Have their blood pressure measured with a non-invasive blood pressure cuff
* Attend 1 focus group (optional)

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Lives, works, or spends much of their time in the South Side of Chicago neighborhood
* Self-reports diagnosis of hypertension or high blood pressure by a clinician
* Endorses elevated depressive symptoms as Patient Health Questionnaire (PHQ)-9 scores ≥10
* Not taking antidepressant medication or stable on antidepressant medication for ≥6 months as self-reported

Exclusion Criteria:

* <18 years old
* Severe mental illness (e.g., bipolar disorder, psychosis)
* Current suicidal ideation (PHQ-9 item 9) or recent (past 6 months) suicide attempt
* Unable to provide informed consent or complete study activities in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness: Depressive Symptom Response | From enrollment to the end of treatment at 8 weeks
  Depressive symptoms are defined as signs and feeling that indicate that a person may be experiencing depression, such as sadness, fatigue, loss of interest or pleasure, and change in appetite. As a clinically sensitive measures of depressive symptom response, participants will complete the Centers for Epidemiologic Studies Depression Scale (CES-D). The CES-D consists of twenty items rated on a four-point Likert scale from 1 (Rarely or None of the time) to 4 (Most or All of the time). Total scores range from 0 to 60, with higher scores indicating a greater burden of depressive symptoms.
  The CES-D is often used in clinical trials and will be used as a measure of effect of the intervention as change in depressive symptoms and has been validated in diverse populations.
Effectiveness: Systolic Blood Pressure Response | From enrollment to the end of treatment at 8 weeks
  Blood pressure (BP) will be measured with an automated BP cuff. Participants will be instructed to rest quietly for 5 minutes, sit upright with feet on the floor, and keep their arm on a flat surface at heart level. Two readings will be taken and averaged. A clinically meaningful change in systolic BP, as defined as a decrease of ≥5 mmHg, would be indicative of a clinical effect of the intervention.
Implementation: Acceptability | Assessed every 6 during the clinical trial enrollment and follow-up for up to 3 years
  One of the primary implementation outcomes will be acceptability of the intervention and its implementation from the perspectives of participants, community members, and organizational leadership. Acceptability will be measured using the Acceptability of Intervention Measure (AIM). The AIM is a 4-item measure with each item scored using a 5-point Likert scale ranging from 1 (Completely disagree) to 5 (Completely agree). AIM scores range from 4 to 20, with higher scores indicating greater acceptability.
Implementation: Appropriateness | Assessed every 6 during the clinical trial enrollment and follow-up for up to 3 years
  One of the primary implementation outcomes will be appropriateness of the intervention and its implementation from the perspectives of participants, community members, and organizational leadership. Appropriateness will be measured using the Intervention Appropriateness Measure (IAM). The IAM is a 4-item measure with each item scored using a 5-point Likert scale ranging from 1 (Completely disagree) to 5 (Completely agree). IAM scores range from 4 to 20, with higher scores indicating greater appropriateness.
Implementation: Feasibility | Assessed every 6 during the clinical trial enrollment and follow-up for up to 3 years
  One of the primary implementation outcomes will be feasibility of the intervention and its implementation from the perspectives of participants, community members, and organizational leadership. Feasibility will be measured using the Feasibility of Intervention Measure (FIM). The FIM is a 4-item measure with each item scored using a 5-point Likert scale ranging from 1 (Completely disagree) to 5 (Completely agree). FIM scores range from 4 to 20, with higher scores indicating greater feasibility.

SECONDARY OUTCOMES:
Effectiveness: Depressive Symptom Remission | From enrollment to the end of treatment at 8 weeks
  Depressive symptoms are defined as signs and feeling that indicate that a person may be experiencing depression, such as sadness, fatigue, loss of interest or pleasure, or change in appetite. As a measure of depression that is commonly used in medical care, participants will complete the Patient Health Questionnaire 9-item scale (PHQ-9). The PHQ-9 consists of 9 items that are rated on a four-point Likert scale from 0 (Not at all) to 3 (Nearly every day). Total scores range from 0 to 27, where higher score indicate greater burden of depressive symptoms. Scores ≥10 on the PHQ-9 are suggestive of a depressive episode.
  The PHQ-9 is consistent with measurement of depressive symptoms in medical/clinical settings and will serve as a clinically meaningful indicator of improvement in depressive symptoms (50% decrease in PHQ-9 score and/or PHQ-9 score <10).
Effectiveness: Blood Pressure Control | From enrollment to the end of treatment at 8 weeks
  Blood pressure control is defined as maintaining blood pressure within a healthy range (i.e., <120/<80 mmHg for healthy adults; <130/<80 mmHg for adults with hypertension). Blood pressure will be measured with an automated BP cuff. Participants will be instructed to rest quietly for 5 minutes, sit upright with feet on the floor, and keep their arm on a flat surface at heart level. Two readings will be taken and averaged.
  Blood pressure control (clinically meaningful indicator) will be defined as <130/<80 mmHg, per American Heart Association guidelines of blood pressure control among individuals diagnosed with hypertension.
Effectiveness: Medication Adherence | From enrollment to the end of treatment at 8 weeks
  Medication adherence is defined as whether a person takes a medication as prescribed (e.g., twice daily). Medication adherence will be measured using the Hill-Bone Compliance to High Blood Pressure Therapy Scale. The Hill-Bone Compliance Scale is a 14-item scale with each item scored using a 4-point Likert scale ranging from 1 (All of the time) to 4 (None of the time). One item is reverse coded. Total scores range from 14 to 56, where higher scores indicate poorer medication adherence.
Implementation: Fidelity | Assessed after each intervention group during the clinical trial enrollment and follow-up for up to 3 years
  Fidelity will be assessed by how well the interventionists, community members, organizational leaders, and researchers adhere to the intervention and implementation protocols. Specifically fidelity to the intervention protocol will be measured using the Mindfulness-Based Interventions: Teaching Assessment Criteria (MBI:TAC). Ratings will be completed by the group leaders (self-ratings) and by trained research team members. The MBI:TAC summary sheet evaluates instructor competency across 6 domains, each comprising 3 to 5 key features. Items are scored using a 6-point Likert scale ranging from 1 (Incompetent) to 6 (Advanced). Total scores range from 27 to 162, with higher scores indicating greater competency in delivering the intervention and, therefore, greater intervention fidelity.

CONTACTS AND LOCATIONS:
Overall Officials: Allison J Carroll, PhD, Principal Investigator — Northwestern University
Locations (1):
- Triedstone Church of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All datasets that can be shared will be deposited in openICPSR, a repository for social, behavioral, and health sciences research data. The participant dataset will include self-reported demographics, psychological metrics, clinical data. The community partners dataset will include coded qualitative responses. The investigators will share de-identified individual-participant level (IPD) data. Item-level data will be shared openly, along with example quantifications and transformations from initial raw data. Final files used to generate specific analyses to answer the Specific Aims and related results will also be shared. Appropriate measures such as removing or recoding identifiers (per Section 164.514(a) of the HIPAA Privacy Rule) will be used for data de-identification and sharing. To facilitate interpretation of the data, data dictionaries, statistical analysis plans, and data collection instruments will be shared and associated with the relevant datasets.
Time Frame: The IPD will be available with the publication of the primary study outcomes.
Access Criteria: All datasets that can be shared will be deposited in openICPSR, a repository for social, behavioral, and health sciences research data. The participant dataset will include self-reported demographics, psychological metrics, clinical data. The community partners dataset will include coded qualitative responses. The investigators will share de-identified individual-participant level (IPD) data. Item-level data will be shared openly, along with example quantifications and transformations from initial raw data.

REFERENCES:
- [Background] Burnett-Zeigler I, Zhou E, Martinez JH, Zumpf K, Lartey L, Moskowitz JT, Wisner KL, McDade T, Brown CH, Gollan J, Ciolino JD, Schauer JM, Petito LC. Comparative effectiveness of a mindfulness-based intervention (M-Body) on depressive symptoms: study protocol of a randomized controlled trial in a Federally Qualified Health Center (FQHC). Trials. 2023 Feb 17;24(1):115. doi: 10.1186/s13063-022-07012-2. PMID 36803835